CLINICAL TRIAL: NCT00245622
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of Subcutaneous Tovaxin in Subjects With CIS or RR-MS
Brief Title: Autologous T Cell Vaccine (TCV) for Multiple Sclerosis
Acronym: TERMS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Opexa Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-00
Record Dates: First submitted 2005-10-20; First posted 2005-10-28 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-02

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Phase 2b Tovaxin; Clinically Isolated Syndrome (CIS); Relapse-Remitting Multiple Sclerosis (RR-MS)
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tovaxin Autologous T cell vaccine (Experimental): 2.0 mL subcutaneous formulated with 30-45 million autologous myelin reactive T cells
  Interventions: Biological: Tovaxin Autologous T cell vaccine
- Placebo (Placebo Comparator): 2.0 mL subcutaneous injections without autologous myelin reactive T cells
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Tovaxin Autologous T cell vaccine — subcutaneous injections administered by healthcare provider at weeks 0, 4, 8, 12, and 24
  Arms: Tovaxin Autologous T cell vaccine
Biological: Placebo — subcutaneous injections administered by healthcare provider at weeks 0, 4, 8, 12, and 24
  Arms: Placebo

SUMMARY:
This is a 1 year study to evaluate the efficacy, safety, and tolerability of Tovaxin T cell therapy in subjects with a clinically isolated syndrome (CIS) and relapse-remitting multiple sclerosis (RR-MS).

DETAILED DESCRIPTION:
A 2 arm, 52 week parallel-group of Tovaxin versus placebo in subjects with CIS or RR-MS. Subjects who provide written, informed consent will complete screening and procurement assessments and provide blood to be used for vaccine production. Eligible subjects will be enrolled to receive either Tovaxin or placebo and will complete baseline assessments. Randomization and enrolled subjects will receive study treatment by subcutaneous injections at weeks 0, 4, 8, 12, and 24. Subjects will be monitored by CBC, serum chemistries, urinalysis, Expanded Disability Status Scale (EDSS), MSFC, MSQLI, magnetic resonance imaging (MRI), and monitor myelin reactive T cells for safety, efficacy, and tolerability of Tovaxin.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 55 years old
* Presence of myelin reactive T cells at screening
* Diagnosis of CIS with screening MRI that fulfils the Barkhof criteria - dissemination in space
* Diagnosis of MS within the past 10 years according to the McDonald criteria (2005)
* Baseline EDSS score between 0 and 5.5 inclusively

Exclusion Criteria:

* Unable to produce T cell vaccine
* Disease-modifying treatment for MS during the last 30 days and 60 days for steroidal treatments
* Diagnosis of progressive-relapsing, secondary progressive, or primary progressive MS
* Planned pregnancy, currently pregnant, or breastfeeding
* Any prior treatment with total lymphoid irradiation, cladribine, T cell or T cell receptor vaccination

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2006-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy, safety, and tolerability of Tovaxin TCV in subjects with CIS or RR-MS | 1 year

SECONDARY OUTCOMES:
To evaluate biomarkers of efficacy of Tovaxin TCV and effects of Tovaxin TCV on epitope spreading | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Edward J Fox, M.D., Ph.D., Study Chair — Central Texas Neurology Consultants; Jaye Thompson, Ph.D., Study Director — Opexa Therapeutics, Inc.
Locations (33):
- United States (33):
  - North Central Neurology Associates, PC, Cullman, Alabama
  - Xenoscience - 21st Century Neurology, Phoenix, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - Alta Bates Summit Medical Center - East Bay Physicians Medical Group, Berkeley, California
  - Patricia A Fodor, PC, Colorado Springs, Colorado
  - Bradenton Neurology, Bradenton, Florida
  - Neurological Associates, Pompano Beach, Florida
  - Lovelace Scientific Resources, Sarasota, Florida
  - Shepherd Center, Atlanta, Georgia
  - Medical College of Georgia - Department of Neurology, Augusta, Georgia
  - Consultants in Neurology, Ltd., Northbrook, Illinois
  - Allied Physicians Inc, Fort Wayne, Indiana
  - MidAmerica Neuroscience Institute, Lenexa, Kansas
  - Associates in Neurology, Lexington, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - Research Nurse Specialists, Lafayette, Louisiana
  - St Mary's of Michigan - Field Neuroscience Institute, Saginaw, Michigan
  - Ayres & Associates Clinical Trials, Lebanon, New Hampshire
  - Upstate Clinical Research, LLC, Albany, New York
  - Winthrop University Hospital - Clinical Trials Unit, Mineola, New York
  - University Hospital and Medical Center Stony Brook New York, Stony Brook, New York
  - Neurology Consultants of the Carolinas, PA, Charlotte, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Neurology & Neuroscience Associates, Inc., Akron, Ohio
  - Neurological Research Institute, Columbus, Ohio
  - Neurology Specialists, Inc, Dayton, Ohio
  - Providence St. Vincent Medical Center - Northwest MS Center, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The Maxine Mesinger MS Clinic/Baylor College of Medicine, Houston, Texas
  - Central Texas Neurology, Round Rock, Texas
  - Integra Clinical Research, LLC, San Antonio, Texas
  - MS Center at Evergreen, Kirkland, Washington
  - Capitol Neurology, Charleston, West Virginia

REFERENCES:
- [Result] Fox E, Markowitz C, Cohan S, Wynn D. TERMS Trial TCV Secondary Analysis of Clinical and Immunological Outcoms in Patients with Relapsing Remitting MS. Poster presentation P06.132 at the 61st Annual Meeting of the American Academy of Neurology (AAN) on 01 May 2009.
- [Derived] Fox E, Wynn D, Cohan S, Rill D, McGuire D, Markowitz C. A randomized clinical trial of autologous T-cell therapy in multiple sclerosis: subset analysis and implications for trial design. Mult Scler. 2012 Jun;18(6):843-52. doi: 10.1177/1352458511428462. Epub 2011 Nov 6. PMID 22065170